CLINICAL TRIAL: NCT02880423
Title: Salpingectomy During Cesarean Section, for Risk Reduction of Ovarian Cancer, Compared With Tubal Ligation- Morbidity and Long Term Complications
Brief Title: Salpingectomy During Cesarean Section
Acronym: SCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, enab.kadour, MD, Bnai Zion Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0012-16BNZ
Record Dates: First submitted 2016-07-29; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: salpingectomy; cesarean section; tubal ligation; morbidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- salpingectomy group I (Other): salpingectomy during cesarean section for sterilization
  Interventions: Procedure: salpingectomy group I
- tubal ligation group II (Active Comparator): tubal ligation in cesarean section
  Interventions: Procedure: tubal ligation group II

INTERVENTIONS:
Procedure: tubal ligation group II — Every woman , who is eligible to enter the study in terms of the above criteria , will receive a detailed explanation of the study and will review the consent form , and then be asked whether she agrees to participate in . If so , the participant will stamped on the informed consent form .
  The control group will be women who undergo tubal ligation method BTL during cesarean section . All women will be invited to follow up about three months after surgery. The women will answer questionnaire to quantify the symptoms of menopause by NAMS , blood test for AMH and sonar and Doppler examination of both the ovaries
  Arms: tubal ligation group II
Procedure: salpingectomy group I — women who agreed to participate in the study and assigned randomly to this group will have salpingectomy during cesarean section for sterilization.
  Arms: salpingectomy group I

SUMMARY:
Based on the accumulated literature, salpingectomy may significantly reduce the risk for ovarian cancer. If investigators can prove that there is no increase in surgical complications and morbidity during salpingectomy in CS, compared to tubal ligation, investigators can recommend for women who are interested in sterilization- salpingectomy during cesarean section .

DETAILED DESCRIPTION:
Until recently, ovarian resection was considered the only option to prevent ovarian cancer. Recently new evidence showing that the fallopian tube itself may be the source of certain types of ovarian cancer. So salpingectomy, may offer some protection. However, the extent of this protection has not been determined. Therefore, and based on the foregoing, the investigators think there is an advantage in removal of fallopian tubes rather than tubal ligation Cesarean sections. Given the lack of evidence in the literature about the complications of this procedure, currently the investigators organize a study examines the rate of complications of salpingectomy compared to tubal ligation during cesarean section.

Therefore, the main objective of the study is to assess the incidence of intra-operative complications during cesarean section.

The effect of the procedure will be examined on the following indicators:

1. The duration of the operation,
2. The rates of bleeding during the operation as estimated by the surgeon,
3. hemoglobin before and after the surgery,
4. Rates of giving blood or after surgery
5. The technical difficulty in performing tubal resection according to surgeon assessment
6. The need for further surgical intervention

A secondary objective of the study is evaluating the long-term complications:

1. Assessment of pain intensity at three months after surgery
2. Evaluation of menopausal symptoms, three months after surgery
3. Test ovarian sonar and Doppler three months after surgery
4. Testing the value of AMH three months after surgery

ELIGIBILITY:
Inclusion Criteria:

* Women planned for cesarean section , according to medical or obstetric indication , and seek sterilization
* Women aged 30 and older
* Women who are capable to understand , read and sign an informed consent form

Exclusion Criteria:

* women aged less then 30 years
* women who disagree to participate in the research

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
intra- operative complications | 5 days
  operation duration,hemorrhage, technical difficulty in performing salpingectomy during CS

SECONDARY OUTCOMES:
long term complication | 3 months
  pain after surgery, signs and symptoms of menopause, reduced ovarian reserve by AMH test

CONTACTS AND LOCATIONS:
Overall Officials: sagi shlomi, md, Study Chair — helsinki bnai zion
Locations (1):
- ISRAEL, Haifa, Israel, Israel

IPD SHARING:
Plan to Share IPD: No